CLINICAL TRIAL: NCT03008642
Title: CO-Rebreathing in Comparison to Isotopic Red Cell Volume Determination in the Diagnosis of Primitive and Secondary Polycythemia: a Multicentric Study. Co-Rebreathing for the Measurement of Total Red Cell Mass in Polycythemia.
Brief Title: CO-Rebreathing in Comparison to Isotopic Red Cell Volume Determination in the Diagnosis of Primitive and Secondary Polycythemia
Acronym: Poly-CO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI2016_843_0032
Record Dates: First submitted 2016-12-01; First posted 2017-01-02 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Polycythemia
Keywords: Polycythemia; CO-Rebreathing; red cell mass determination; myeloproliferative neoplasms
MeSH Terms: conditions — Polycythemia; Myeloproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CO-Rebreathing (Experimental): The intervention consists in one red cell mass determination using the CO-Rebreathing technique at diagnosis of polycythemia, in addition to the regular tests performed in this indication, including RCM isotopic measurement.
  Interventions: Other: CO-Rebreathing technique at diagnosis of polycythemia

INTERVENTIONS:
Other: CO-Rebreathing technique at diagnosis of polycythemia — The intervention consists in one red cell mass determination using the CO-Rebreathing technique at diagnosis of polycythemia, in addition to the regular tests performed in this indication, including RCM isotopic measurement.

SUMMARY:
The optimized CO-Rebreathing is an efficient method to evaluate the red cell mass and has been used in the vast majority of studies in sport medicine. However, this method has never been evaluated on a large scale in the diagnosis of primitive or secondary polycythemia. The standard procedure to evaluate the red cell mass is based on isotopic measurement using Cr51-labelled red cells, but its lack of availability in many centers highlights the need for a non-invasive and rapid alternative method. The purpose of this study is to evaluate and validate the CO-Rebreathing method in this set of indications.

DETAILED DESCRIPTION:
The definition of a true polycythemia is stricto sensu an increased red cell mass (RCM) above 125% of the expected value depending on the size and the weight of the patient. However, this measurement requires an isotopic labeling of red cells and is not available in most of the hospitals. Therefore, the diagnosis of polycythemia, and particularly Polycythemia Vera (PV) is based on routine red blood cells parameters, i.e. hemoglobin level and hematocrit. If these parameters are efficient in marked polycythemia, discrepancies have been observed in milder cases. Two situations where a RCM evaluation is particularly required can be described:

* In patients with a hematocrit level between 52 and 60% (men) or between 48 and 56% (women) in order to limit invasive investigations to patients with a confirmed polycythemia diagnosis
* In JAK2V617F positive myeloproliferative neoplasms (MPN) with hematocrit and hemoglobin levels under the PV cut-off in order to discriminate between masked PV and essential thrombocythemia CO-Rebreathing is a fast, non invasive alternative method for RCM evaluation. It is based on the high affinity of carbon monoxide (CO) for hemoglobin. The decrease in the HbCO percentage after CO inhalation is dependent on the total hemoglobin mass from which RCM can be obtained. The investigators propose a tri-centric study evaluating CO-Rebreathing as an alternative tool to measure RCM in the diagnosis of polycythemia in the two categories of patients described above.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient
2. Informed consent obtained
3. Requirement of an isotopic red cell mass determination:

   a - Hematocrit between 52 and 60% (men) or 48 and 56% (women) with no argument for a PV (JAK2V617F negative, EPO level normal/high).

   b - Patients with a JAK2V617F positive MPN and a hematocrit level between 46 and 50% (women) or 48 and 52% for men.
4. No recent vascular event (<6 mois)
5. No unstable coronaropathy
6. Non smoking since 24 hours.
7. ECOG <2
8. Negativity of pregnancy test/effective contraception for childbearing age women,
9. Health insurance

Exclusion Criteria:

1. Recent venous event <1 months, cerebral stroke < 6 mois)
2. Evolutive cardiopathy (< 6 months)
3. Chronic Respiratory failure
4. Smokers with no withdrawal in the last 24 hours before CO-Rebreathing
5. Basal HbCO>7% the day of CO-Rebreathing
6. Pregnant or breast feeding women
7. Patient enable to give an informed consent
8. Inclusion in an interventional clinical trial in the last three months.
9. Any contraindication to lung function testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
equivalence of RCM determination by CO-Rebreathing in comparison to the traditional isotopic measurement in the diagnosis of polycythemia | 1 month
  The primary outcome is to prove the equivalence of RCM determination by CO-Rebreathing in comparison to the traditional isotopic measurement in the diagnosis of polycythemia.

SECONDARY OUTCOMES:
AE / SAE / EI | 1 month
  Incidence, grade type according to NCI-CTCAE v4.0
Cumulative incidence of thrombotic and hemorrhagic complications | 1 month
  Cumulative incidence of thrombotic and hemorrhagic complications List according to PT1 protocol.
Deaths and causes | 1 month
  Deaths and causes
Analysis of the results of VGTCO and VGTi | 1 month
  Analysis of the results of VGTCO and VGTi as a function of hemoglobin and hematocrit

CONTACTS AND LOCATIONS:
Overall Officials: Loïc GARCON, professor, Study Director — CHU Amiens-Picardie; Lydia ROY, Doctor, Principal Investigator — CHU Henri Mondor, France; Marjolaine GEORGES, Doctor, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

REFERENCES:
- [Result] Maaziz N, Georges M, Basille D, Gallet M, Gardie B, Diouf M, Garcon L, Girodon F. Carbon monoxide rebreathing method is a reliable test to evaluate the red cell mass in polycythaemia. Br J Haematol. 2024 Feb;204(2):706-709. doi: 10.1111/bjh.19169. Epub 2023 Dec 3. No abstract available. PMID 38044575